CLINICAL TRIAL: NCT07145073
Title: Repetitive Transcranial Alternating Current Stimulation(rtACS) for the Treatment of Optic Neuropathies
Brief Title: Repetitive Transcranial Alternating Current Stimulation (rtACS) for the Treatment of Optic Neuropathies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202409124DSE
Record Dates: First submitted 2025-08-11; First posted 2025-08-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma
Keywords: Glaucoma; electrical stimulation
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repetitive Transcranial Alternating Current Stimulation treatment (Experimental): Participants will receive 10 days of repeated transcranial alternating current stimulation in hospital.
  Interventions: Device: DC-Stimulator MC
- Sham Repetitive Transcranial Alternating Current Stimulation (Sham Comparator): Participants will receive 10 days of repeated transcranial alternating current stimulation treatment (no active stimulation) in hospital.
  Interventions: Device: DC-Stimulator MC

INTERVENTIONS:
Device: DC-Stimulator MC — Experimental：Participants will receive 10 days of repeated transcranial alternating current stimulation treatment in hospital.
  Arms: Repetitive Transcranial Alternating Current Stimulation treatment
Device: DC-Stimulator MC — Sham Comparator：Participants will receive 10 days of repeated transcranial alternating current stimulation treatment (no active stimulation) in hospital.
  Arms: Sham Repetitive Transcranial Alternating Current Stimulation

SUMMARY:
The goal of this study is to see whether repeated transcranial alternating current stimulation can activate impaired retinal ganglion cells and improve both structural and functional outcomes in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18.
2. Clinical diagnosis of glaucoma, with Humphrey Visual Field 24-2 mean deviation (MD) between -22 dB and -5 dB, and Visual Field Index (VFI) between 10% and 90%. The visual field test at screening must meet the following reliability indices:

   * Fixation losses (FL) ≤ 33%
   * False-negative rate (FNR) ≤ 20%
   * False-positive rate (FPR) ≤ 20% At initial screening, the difference in MD between two consecutive visual field tests must be less than 2 dB.
3. Best-corrected visual acuity (BCVA) ≥ 0.2 in the worse eye selected for stimulation treatment.
4. If a participant has two eyes meeting study criteria, one eye will be randomly selected by computer for study participation.
5. In the opinion of the investigator the participant's eye pressure must be clinically stable.
6. Participant must has the ability to comply with the requirements of the study and complete the schedule of events.
7. Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.
8. Optical coherence tomography (OCT) imaging shows measurable changes in either peripapillary retinal nerve fiber layer (RNFL) thickness or macular ganglion cell-inner plexiform layer thickness.

Exclusion Criteria:

1. History of ocular herpes.
2. Pathological nystagmus.
3. Retinal disease sufficient to affect vision.
4. Corneal opacity affecting vision.
5. Cataract affecting vision.
6. Uveitis or other intraocular inflammatory disease.
7. Implanted electronic devices such as a pacemaker.
8. Rheumatologic or autoimmune disease.
9. Brain tumor or intracranial magnetic metallic implants.
10. History of epilepsy.
11. Periocular skin lesions.
12. Anxiety with Geriatric Anxiety Scale score > 12.
13. History of claustrophobia.
14. Participation in another clinical trial within the past 3 months involving medication or training that could affect the eyes.
15. Physical or mental conditions that may increase the risk of participation or interfere with study assessments (e.g., dementia).
16. Previous ocular electrical stimulation treatment or visual training study within the past 12 months.
17. Uncontrolled hypertension or diabetes.
18. Pregnant or breastfeeding.
19. History of craniotomy, burr hole surgery, head trauma, intracranial tumor, vascular malformation, or intracranial surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in visual field mean deviation (MD) from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Visual field testing will be performed with the Humphrey field analyzer

SECONDARY OUTCOMES:
Change in visual field mean deviation (MD) from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Visual field testing will be performed with the Humphrey field analyzer
Change in visual field mean deviation (MD) from baseline to post-treatment | From treatment initiation to 19 days after treatment initiation
  Visual field testing will be performed with the Humphrey field analyzer
Change in visual field mean deviation (MD) from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Visual field testing will be performed with the Humphrey field analyzer
Change in sensitivity at each of the 52 test points in the 24-2 visual field from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
Change in targeted mean deviation from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
Change in targeted mean deviation from baseline to post-treatment | From treatment initiation to 19 days after treatment initiation
Change in targeted mean deviation from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
Change in targeted mean deviation from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
Visual function analysis from baseline to post-treatment | From treatment initiation to 5 days after treatment initiation
  Visual acuity measured by Landolt C Chart.
Visual function analysis from baseline to post-treatment | From treatment initiation to 5 days after treatment initiation
  Contrast sensitivity measured by CSV-1000
Visual function analysis from baseline to post-treatment | From treatment initiation to 5 days after treatment initiation
  Contrast sensitivity measured by Pelli-Robson Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 5 days after treatment initiation
  Contrast sensitivity measured by MARS Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 5 days after treatment initiation
  Color vision measured by HRR pseudoisochromatic test
Visual function analysis from baseline to post-treatment | From treatment initiation to 5 days after treatment initiation
  Continuous Chinese reading acuity measured by Paragraph Chinese Reading Acuity Test (P-CRAT)
Visual function analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Visual acuity measured by Landolt C Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Contrast sensitivity measured by CSV-1000
Visual function analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Contrast sensitivity measured by Pelli-Robson Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Contrast sensitivity measured by MARS Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Color vision measured by HRR pseudoisochromatic test
Visual function analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation]
  Continuous Chinese reading acuity measured by Paragraph Chinese Reading Acuity Test (P-CRAT)
Visual function analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Visual acuity measured by Landolt C Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Contrast sensitivity measured by CSV-1000
Visual function analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Contrast sensitivity measured by Pelli-Robson Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Contrast sensitivity measured by MARS Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Color vision measured by HRR pseudoisochromatic test
Visual function analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Continuous Chinese reading acuity measured by Paragraph Chinese Reading Acuity Test (P-CRAT)
Visual function analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Visual acuity measured by Landolt C Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Contrast sensitivity measured by CSV-1000
Visual function analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Contrast sensitivity measured by Pelli-Robson Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Contrast sensitivity measured by MARS Contrast Sensitivity Chart
Visual function analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Color vision measured by HRR pseudoisochromatic test
Visual function analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Continuous Chinese reading acuity measured by Paragraph Chinese Reading Acuity Test (P-CRAT)
Quality of life analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Vision-related quality of life assessed using the National Eye Institute 25-Item Visual Function Questionnaire (NEI VFQ-25). Scores are converted to a 0-100 scale, where higher scores indicate better vision-related quality of life.
Quality of life analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Health status assessed using the 36-Item Short Form Health Survey (SF-36). Scores for each domain and the overall score range from 0 to 100, where higher scores indicate better health status.
Quality of life analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Mobility in daily life assessed using the Mobility questionnaire. This questionnaire focuses on difficulties related to mobility and driving. Scores are reported on a 0-172 scale, where higher scores indicate greater difficulty with mobility and driving in daily life.
Quality of life analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Vision-related quality of life assessed using the National Eye Institute 25-Item Visual Function Questionnaire (NEI VFQ-25). Scores are converted to a 0-100 scale, where higher scores indicate better vision-related quality of life.
Quality of life analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Health status assessed using the 36-Item Short Form Health Survey (SF-36). Scores for each domain and the overall score range from 0 to 100, where higher scores indicate better health status.
Quality of life analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Mobility in daily life assessed using the Mobility questionnaire. This questionnaire focuses on difficulties related to mobility and driving. Scores are reported on a 0-172 scale, where higher scores indicate greater difficulty with mobility and driving in daily life.
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Peripapillary retinal nerve fiber layer (RNFL) thickness (μm)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Macular ganglion cell-inner plexiform layer thickness (μm)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Optic nerve head cup-to-disc ratio (%)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Peripapillary retinal nerve fiber layer (RNFL) thickness (μm)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Macular ganglion cell-inner plexiform layer thickness (μm)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Optic nerve head cup-to-disc ratio (%)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Peripapillary retinal nerve fiber layer (RNFL) thickness (μm)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Macular ganglion cell-inner plexiform layer thickness (μm)
Optical coherence tomography (OCT) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Optic nerve head cup-to-disc ratio (%)
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Peripapillary vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  capillary density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Superficial density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  deep density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  foveal vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  parafoveal vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 12 days after treatment initiation
  Foveal avascular zone (FAZ)
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Peripapillary vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  capillary density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Superficial density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  deep density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  foveal vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  parafoveal vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 26 days after treatment initiation
  Foveal avascular zone (FAZ)
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Peripapillary vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  capillary density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Superficial density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  deep density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  foveal vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  parafoveal vessel density
Optical coherence tomography angiography(OCT-A) analysis from baseline to post-treatment | From treatment initiation to 166 days after treatment initiation
  Foveal avascular zone (FAZ)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Hawaii, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided